CLINICAL TRIAL: NCT06526676
Title: Clinical Outcomes and Predictors of Major Adverse Events in Patients Treated for Juxtarenal, Pararenal and Thoracoabdominal Aortic Aneurysms With Physician-Modified Fenestrated and Branched Stent Grafts
Brief Title: Clinical Outcomes and Major Adverse Events in Patients Treated With Physician-Modified Fenestrated and Branched Stent Grafts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Bernardo Mendes, MD, Principal Investigator, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-1031
Record Dates: First submitted 2024-06-03; First posted 2024-07-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Juxtarenal Aortic Aneurysm; Pararenal Aneurysm; Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Subjects with short neck infrarenal, juxtarenal, suprarenal and extent IV TAA (Experimental): Subjects will have their aortic aneurysms repaired using an investigational physician-modified graft
  Interventions: Device: Cook Alpha TX2 Stent Graft, Cook Zenith TX2, and Cook Zenith Fenestrated Stent Graft
- Subjects with thoracoabdominal aortic aneurysms (Experimental): Subjects will have their aortic aneurysms repaired using an investigational physician-modified graft
  Interventions: Device: Cook Alpha TX2 Stent Graft, Cook Zenith TX2, and Cook Zenith Fenestrated Stent Graft
- Subjects with urgent or emergent aneurysms (Experimental): Subjects will have their aortic aneurysms repaired using an investigational physician-modified graft
  Interventions: Device: Cook Alpha TX2 Stent Graft, Cook Zenith TX2, and Cook Zenith Fenestrated Stent Graft

INTERVENTIONS:
Device: Cook Alpha TX2 Stent Graft, Cook Zenith TX2, and Cook Zenith Fenestrated Stent Graft — Physician-modified stent grafts that utilizes multiple stent grafts with a combination of fenestrations and/or branches

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of endovascular treatment of juxtarenal, pararenal and thoracoabdominal aortic aneurysms (with or without iliac artery involvement) using physician-modified stent grafts with a combination of fenestrations and/or branches.

ELIGIBILITY:
Inclusion Criteria:

A patient may be included in the study if at least one of the following is present and is considered appropriate for treatment with a physician modified stent graft. Patients must be deemed high risk for traditional open surgical repair, if any of the following conditions are present.

Patients will be deemed physiologically high risk if any of the following conditions are present:

* Older than 75 years of age
* Chronic obstructive pulmonary disease
* Congestive heart failure
* Previous myocardial infarction, coronary stent, or bypass
* Chronic renal insufficiency with baseline eGFR < 40 ml/min
* American Society of Anesthesiologist (ASA) score > 3

Patient will be deemed anatomically high risk if any of the following conditions are present:

* Prior intraabdominal operation(s)
* Prior abdominal wall reconstructions. (ie. Ventral hernia repairs)
* Prior radiation therapy targeting abdomen and/or pelvis
* History of intraabdominal sepsis. (ie. Diverticulitis managed with percutaneous drainage)

Patients will then be included in one of three arms with the inclusion criteria specified as follows:

* Arm 1 (Short neck infrarenal, juxtarenal, suprarenal and extent IV TAA)

  * Juxtarenal, pararenal, suprarenal or extent IV thoracoabdominal aortic aneurysm or dissection with a diameter ≥ 5.5 cm or 2 times the normal aortic diameter.
  * Juxtarenal, pararenal, suprarenal or extent IV thoracoabdominal aneurysm with a history of growth ≥ 0.5 cm in one year.
  * Juxtarenal, pararenal, suprarenal or extent IV thoracoabdominal saccular aneurysms deemed at significant risk for rupture based upon physician interpretation.
  * Presence of juxtarenal, pararenal, suprarenal or extent IV thoracoabdominal aortic aneurysm not meeting one of the above-mentioned criteria with or without unilateral or bilateral common iliac artery aneurysm with diameter ≥ 3.5-cm or saccular morphology with no suitable landing zone proximal to iliac bifurcation.
* Arm 2 (Thoracoabdominal aortic aneurysms)

  * Extent I, II, or III thoracoabdominal aortic aneurysm or dissection with a diameter ≥ 5.5 cm or 2 times the normal aortic diameter.
  * Extent I, II, or III thoracoabdominal aortic aneurysm with a history of growth ≥ 0.5 cm in one year.
  * Extent I, II, or III thoracoabdominal saccular aortic aneurysms deemed at significant risk for rupture based upon physician interpretation.
  * Presence of Extent I, II, or III thoracoabdominal aortic aneurysm not meeting one of the above-mentioned criteria with or without unilateral or bilateral common iliac artery aneurysm with diameter ≥ 3.5-cm or saccular morphology with no suitable landing zone proximal to iliac bifurcation.
* Arm 3 (Urgent or emergent aneurysms) o Ruptured, contained ruptured or symptomatic juxtarenal, pararenal, suprarenal or thoracoabdominal aortic aneurysm planned to receive urgent or emergent repair within 48 hours of clinical encounter, in patients able to provide informed consent and deemed not a reasonable candidate for open surgery or repair with any commercially available device.

Exclusion Criteria:

Patients must be excluded from the study if any of the following conditions are true:

* Less than 18 years of age
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent by the patient or a legally authorized representative
* Pregnant or breastfeeding
* Life expectancy < 2-years
* Prior open surgical or interventional procedure within 30 days of the anticipated date of the fenestrated-branched procedure, with the exception of planned staged procedures to provide access for repair (e.g. staged iliac conduit, cervical debranching, elephant trunk repair), to facilitate the procedure by allowing open revascularization of a target artery not amenable to revascularization with the investigational device, such as an internal iliac artery, subclavian artery or visceral artery with early bifurcation, tortuosity or occlusive disease preventing successful placement of alignment side stents.
* Patients eligible for treatment with any FDA-approved marketed device within its instructions for use
* Can enroll in a manufacturer-sponsored clinical study at our institution or is willing and eligible to participate in a study with a manufactured-made device at another institution
* Participation in another investigational clinical or device trial, with the exception of participation in another investigational endovascular stent-graft protocol, percutaneous aortic valve protocol, or concomitant clinical trials designed to evaluate medical therapy strategies to reduce perioperative risk during fenestrated-branched endovascular repair, including risks of renal dysfunction, contrast-induced nephropathy, neurologic, spinal cord or cardiac complications, and/or use of advanced imaging to reduce radiation exposure during implantation of these devices. Participation in investigational device trials not encompassed by the IDE protocol should be performed remotely from the fenestrated procedure (>30 days). Examples include remote (>30 days) participation in a thoracic, abdominal, or iliac branch device trial, or participation in a percutaneous aortic valve trial. Participation in medical therapy trial or advanced imaging trial designed to improve peri-operative outcomes or to reduce radiation exposure of fenestrated-branched endografts may be concurrent with the IDE study. Examples include therapy directed to reduce rates of spinal cord injury, stroke and contrast-induced nephropathy associated with implantation of fenestrated-branched stent-grafts or advanced imaging trials designed to reduce radiation exposure during repair.

Medical Exclusion Criteria:

* Known sensitivities or allergies to stainless steel, nitinol, polyester, solder (tin, silver), polypropylene, PTFE, urethane, or gold.
* History of anaphylactic reaction to contrast material that cannot be adequately pre-medicated.
* Uncorrectable coagulopathy.
* Mycotic aneurysm or patients with evidence of active systemic infection.
* History of connective tissue disorder (e.g vascular Ehlers Danlos, Marfan's syndrome), except for those patients who had prior open surgical aortic replacement, where a surgical graft would serve as landing zone for the investigational stent-graft, those who are deemed prohibitive risk for open surgical repair or connective tissue disorders with no effect of vascular system (e.g non-vascular Ehlers Danlos).
* Body habitus that would inhibit X-ray visualization of the aorta and its branches.

Anatomic Exclusion Criteria

* Inadequate femoral or iliac access compatible with the required delivery systems.
* Inability to perform a temporary or permanent open surgical or endovascular iliac conduit for patients with inadequate femoral/iliac access.
* Absence of a non-aneurysmal aortic segment in the distal thoracic aorta above the diaphragmatic hiatus with:

  * A diameter measured outer wall to outer wall of no greater than 42mm and no less than 21 mm;
  * Parallel aortic wall with <20% diameter change and without significant calcification and/or thrombus in the selected area of seal zone
* Visceral vessel anatomy not compatible with fenestrated/branched stent graft visceral vessel incorporation due to excessive occlusive disease or small size not amenable to stent graft placement
* Unsuitable distal iliac artery fixation site and anatomy for iliac limb extension or iliac branch device as per devices' instructions for use (IFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with major adverse events | 30 days
  Total number of patients to experience a major adverse event as defined as any cause mortality, bowel ischemia (requiring surgical therapy), type I myocardial infarction (rise of troponin levels at least 1 value above 99th percentile of upper limit and with at least one of the following: symptoms of acute myocardial ischemia, new ischemic ECG changes, development of new pathological Q waves, imaging evidence of loss of viable myocardium or new regional wall motion abnormalities, or identification of coronary thrombus by angiography or by autopsy), paraplegia (Level 3), renal failure (need for renal replacement therapy or > 50% decline in eGFR), respiratory failure (respiratory failure requiring ventilatory support > 24 hours or re-intubation), major stroke.
Treatment success | 12 months
  Total number of patients to achieve treatment success as defined by: technical success, defined as successful delivery, deployment and withdrawal of the physician-modified endovascular graft with preservation and patency of those branch vessels intended to be preserved; freedom from aneurysm enlargement >5 mm; freedom from secondary interventions for type I or type III endoleak, stent-graft migration, device integrity failure (e. g., fracture), and patency-related events; and freedom from aneurysm rupture or conversion to open repair.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 30 days, 6 months, and annually at 1, 2, 3, 4 and 5 years
  The Short Form Health Survey (SF-36) is a 36-item, participant-reported survey that measures patient health and disability. Possible scores range from 0 to 100, with 0 indicating maximum disability, and 100 indicating no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo C Mendes, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No